CLINICAL TRIAL: NCT06024057
Title: An Expanded Clinical Study Evaluating the AAV2-RPE65 Gene Therapy (LX101) in Patients With Leber's Congenital Amaurosis (LCA)
Brief Title: An Expanded Clinical Study Evaluating the AAV2-RPE65 Gene Therapy(LX101) in Patients With LCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Assessor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX101-EX
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: To Evaluate the Scaling Clinical Study of AAV2-RPE65 Gene Therapy Agent (LX101) in Patients With Congenital Amaurosis (LCA)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LX101 (Experimental)
  Interventions: Drug: LX101

INTERVENTIONS:
Drug: LX101 — LX101 (Containing recombinant human adeno-associated virus serotype 2, AAV2-RPE65 encoding human RPE65 gene).Specification: 0.2mL/bottle.Route of administration: subretinal injection, injection volume 0.3 mL/ eye

SUMMARY:
To evaluate the scaling clinical trail of AAV2-RPE65 gene therapy agent (LX101) in patients with congenital amaurosis (LCA).

DETAILED DESCRIPTION:
This study evaluated the overall safety and initial efficacy of RPE65 mutant congenital amaurosis (RPE65-LCA) in subjects treated with a single, subretinal injection of LX101 (containing recombinant human adeno-associated virus serotype 2, AAV2-RPE65) in the second eye 1 year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Participants in the main study "Exploratory clinical study evaluating AAV2-RPE65 gene therapy formulation (LX101) in patients with congenital amaurosis (LCA) 2) Willingness to participate in the extended study, subject and/or their guardian signing a written informed consent and complying with a long-term follow-up protocol

Exclusion Criteria:

* Have any of the following eye conditions:

  1. Subjects with SAE in the "Exploratory clinical Study Evaluating AAV2-RPE65 gene therapy agent (LX101) in patients with congenital Amaurosis (LCA)
  2. pre-existing eye conditions (such as glaucoma, cornea, or severe lens opacity) that the investigator determines may interfere with planned surgery or with interpretation of the study endpoint;
  3. Screening subjects who had undergone any internal eye surgery in the six months prior to the visit;
  4. Inability or unwillingness to meet the requirements of the study;

Have any of the following systemic conditions:

6) Known allergy to the drug planned for use in the study; 7) Have a history of surgical operations within 1 month before enrollment, and/or present unhealed wounds, ulcers, fractures, etc.; Present infectious disease requiring oral, intramuscular or intravenous administration; 8) Baseline laboratory values for complex systemic diseases or clinically significant abnormalities; 9) Complex systemic diseases include diseases in which the disease itself or the treatment of the disease can alter eye function. For example, the treatment of malignant tumors can affect central nervous system function (e.g., orbital radiation therapy; Leukemia with central/optic nerve involvement); 10) Subjects with a history of immune-damaging diseases due to the possibility of opportunistic infection (e.g., CMV retinitis); Subjects with diabetes or sickle cell disease will be excluded if they have any manifestations of advanced retinopathy, such as macular edema or proliferative changes. Subjects with juvenile rheumatoid arthritis have an increased risk of infection due to poor postoperative wound healing; 11) Participants who cannot discontinue Viagra (Sildenafil) or related compounds used to treat erectile dysfunction during the study period; 12) Subjects who cannot discontinue hydroxychloroquine, Chloroquine, meralide, or any related retinal toxic compound during the study; 13) Any other conditions in which the potential subject is not allowed to complete a follow-up examination during the study, and the investigator believes that there are conditions that make the potential subject unfit for the study.

Fertile subjects with any of the following conditions:

14) Those who do not use effective contraceptive measures; 15) Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2038-09-30 (Estimated)

PRIMARY OUTCOMES:
Local and systemic safety assessment | 52（+4）weeks
  Eye and non-eye adverse events

IPD SHARING:
Plan to Share IPD: No